CLINICAL TRIAL: NCT04396483
Title: Dysfunctional Uterine Bleeding After Tubal Sterilization and Salpingectomy
Brief Title: Dysfunctional Uterine Bleeding After Tubal Sterilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DUBATS
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Contraception; Dysfunctional Uterine Bleeding
Keywords: Dysfunctional uterine bleeding; Tubal sterilization; Salpingectomy; Cesarean section
MeSH Terms: conditions — Metrorrhagia | interventions — Salpingectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubal sterilization "Pomeroy's method" (Experimental)
  Interventions: Procedure: Pomeroy's tubal sterilization
- Salpingectomy (Active Comparator)
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Pomeroy's tubal sterilization — Both Fallopian tubes will be grasped by allis forceps and a kokher forceps will be applied below the allis forceps then excision of tubal part above kokher and transfixation of both ends away from each other during cesarean section
  Arms: Tubal sterilization "Pomeroy's method"
Procedure: Salpingectomy — Both fallopian tubes will be completely removed during cesarean section
  Arms: Salpingectomy

SUMMARY:
In this study, the investigators will compare the frequency and amount of bleeding after tubal sterilization and salpingectomy

DETAILED DESCRIPTION:
Dysfunctional uterine bleeding is common after tubal sterilization.

The investigators will compare the frequency and amount of bleeding after two techniques eithe tubal sterilization by pomeroy's method during cesarean section or complete salpingectomy

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* Patient completed her family
* Patient on cesarean delivery

Exclusion Criteria:

* Tubal sterilization by other methods
* Salpingectomy by laparoscopy
* Patient wishing fertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Dysfunctional bleeding | 1 year after cesarean section
  percentage of cases suffering of dysfunctional bleeding
Amount of bleeding | 1 year after cesarean section
  number of sanitary pads during bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Adel Elgergawy, Tanta, Gharbia Governorate
  - Ayman Shehata Dawood, Tanta, Gharbia Governorate

IPD SHARING:
Plan to Share IPD: Yes
When valid request is present
Supporting Information: Study Protocol
Time Frame: 6 months